CLINICAL TRIAL: NCT04871464
Title: Role and Mechanism of Bifidobacterium Triple Viable Capsules in Improving Motor Symptoms in Patients With Mild to Moderate Parkinson's Disease: a Multicenter Randomized Clinical Study
Brief Title: Role and Mechanism of Probiotics in Improving Motor Symptoms in Mild to Moderate Parkinson's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Houzhen Tuo, Vice-Director of Neurology, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-P2-153-02
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease; Parkinsonian Disorders; Basal Ganglia Diseases; Brain Diseases; Movement Disorders; Neurodegenerative Diseases; Central Nervous System Diseases; Nervous System Diseases
Keywords: Parkinson's disease; Probiotics
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Basal Ganglia Diseases; Brain Diseases; Movement Disorders; Neurodegenerative Diseases; Central Nervous System Diseases; Nervous System Diseases | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Study is double blind design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotics (Experimental): Bifidobacterium triple viable capsules（BIFICO），containing Bifidobacterium longum, Lactobacillus acidophilus and Enterococcus faecalis(each ≥ 1.0×10^7 CFU/capsule)，Day 1-14, 2 capsules twice daily; Day 15-24 weeks, 4 capsules twice daily, taken orally half an hour after meals.
  Interventions: Drug: Live Combined Bifidobacterium,Lactobacillus and Enterococcus Capsules
- Placebo (Placebo Comparator): Placebo，day 1-14, 2 capsules twice daily; Day 15-24 weeks, 4 capsules twice daily, taken orally half an hour after meals.
  Interventions: Other: Placebo
- Healthy control (No Intervention): Healthy subjects without constipation matched for age and sex to PD subjects

INTERVENTIONS:
Drug: Live Combined Bifidobacterium,Lactobacillus and Enterococcus Capsules — Oral
  Other Names: BIFICO
  Arms: Probiotics
Other: Placebo — Oral
  Arms: Placebo

SUMMARY:
This study is a multicenter randomized double-blind placebo-controlled study. The research content is 1. The improvement effect of Bifidobacterium triple viable capsules（BIFICO） on motor symptoms and constipation and sleep in mild to moderate Parkinson's disease and the safety of the study; 2. the mechanism of the improvement effect of intestinal microecological changes on motor and constipation symptoms in mild to moderate Parkinson's disease.

DETAILED DESCRIPTION:
This was a multicenter randomized double-blind placebo-controlled study that included 240 patients with primary PD with modified H-Y stage 1-3, randomly divided into treatment and placebo control groups; On the basis of the original PD medication, the treatment group was given bifidobacterium triple viable capsules (BIFICO) and the control group was given placebo; Patients who met the diagnosis of constipation were given Macrogol 4000 powder and /or Enema glycerine as a rescue medicine, and the observation period was 12+12 weeks.

All subjects underwent the World Movement Disorders Society Parkinson's Disease Comprehensive Rating Scale (MDS-UPDRS), Rome IV Constipation Diagnostic Scale, Cleveland Rating Scale, Parkinson's Disease Sleep Scale-2 (PDSS-2), and General Clinical Outcome Inventory (CGI) scores before and after treatment, and also recorded the patients' single bowel movement time and the use of Macrogol 4000 powder and Enema glycerine , to investigate the improvement effect of Bifido on motor symptoms and non-motor symptoms in PD patients. For the above patients, stool and blood samples were collected at the time of enrollment and at 12 weeks of observation.

At the same time,120 age-and gender-matched healthy adults without constipation were recruited, and their stool and blood samples were collected; the stool samples of PD patients before and after treatment and healthy controls were subjected to the determination of fecal flora 16S DNA abundance. Stool samples of 10 PD patients and 10 healthy controls were taken from each group for metagenomic sequencing. Detection of small molecule metabolites, PD-related genes in blood. To investigate the effect of BIFICO on levodopa pharmacokinetics, levodopa pharmacokinetic measurements will be performed at Friendship Hospital. For patients who agree to participate and sign the informed consent form, blood specimens will be collected consecutively at Visit 2 and Visit 11 after taking Levodopa and Benserazide Hydrochloride Tablets for levodopa blood concentration measurement.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-85 years old, both male and female;
* Patients with primary Parkinson's disease who meet the 2015 MDS clinical diagnostic criteria; PD with modified Hoehn-Yahr stage 1-3 and MDS-UPDRS II+III score ≥ 14 and no significant off periods or off periods ≤ 1.5 hours per day (excluding morning motor inability);
* Pre-enrollment therapeutic medications included Levodopa complex preparation, and all Parkinson's disease medications were unadjusted and motor symptoms were stable for 28 days prior to enrollment;
* No probiotic or/and prebiotic (including lactulose) and antibiotic therapy for 60 days prior to enrollment, and if so, a 60-day washout period;
* Understand and agree to follow the study protocol, agree to be enrolled and sign the informed consent form.

Exclusion Criteria:

* Parkinson's superimposed syndrome and secondary Parkinson's syndrome, such as multiple system atrophy, progressive supranuclear palsy, etc.；
* Taking any probiotic or prebiotic (including lactulose) within 60 days prior to enrollment; having inflammation at any site and using any antibiotic within 60 days prior to enrollment; or having blood leukocytes above the upper limit of normal at screening；
* Combined endocrine disorders, such as history of diabetes or fasting glucose ≥ 7.8 mmol/L;
* Comorbid other neurological disorders, such as cognitive impairment, Mini-Mental State Examination （MMSE） scale score <24; severe anxiety states and/or severe depressive states (Hamilton Depression Inventory-17 item score >17, Hamilton Anxiety Scale score ≥14, or being treated with antidepressant anxiety medication); Note: Those who were taking antidepressant and anxiety drugs and had no adjustment in the last 28 days, and whose score of Hamilton Depression Scale -17 was less than 17, and Hamilton Anxiety Scale score was less than 14 were not included in the exclusion criteria; Severe autonomic nervous disease occurs within 5 years of onset, malignancy, spinal cord lesions, epilepsy, autonomic disorders (urinary retention, urinary incontinence, or upright hypotension , blood pressure drop ≥30/15 mmHg at any time point within 5 minutes of uprightness), etc.; new cerebrovascular disease or sequelae of severe cerebrovascular disease within 6 months, which affects the assessment；
* Gastrointestinal tumors, history of inflammatory bowel disease, other acute and chronic inflammation of the gastrointestinal tract (including acute attacks of cholecystitis) within 3 months；
* History of gastrointestinal surgery (excluding endoscopic resection of gastrointestinal benign polyps, appendicitis resection) or constipation caused by surgery；
* History of anal fissure, perianal abscess, irreversible anal prolapse, pelvic trauma；
* Severe cardiovascular disease (such as congestive heart failure with a heart function classification of Ⅲ-Ⅳ by the American Heart Association, a history of myocardial infarction within 6 months, etc.);
* Severe liver and kidney dysfunction with glutamate-pyruvate transaminase, aspartate transaminase and total bilirubin 2.0 times higher than the upper limit of normal; serum creatinine 2.0 times higher than the upper limit of normal;
* Pregnant and lactating women or women of childbearing age (40-60 years) who are human chorionic gonadotropin (HCG)-positive;
* Known allergy to test drugs or related products;
* People with a history of drug abuse or alcohol dependence;
* Those who have participated in other clinical trials within 3 months prior to enrollment;
* Refusal to enroll and inability to cooperate with the investigator; patients judged by the investigator to be unsuitable for enrollment.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale(MDS-UPDRS)Ⅱ+Ⅲ | 12 weeks
  Part Ⅱ：This measures the motor aspects of activity of daily living and consists of 13 items with scores between 0- 52. Part Ⅲ：This measures the severity of motor symptoms using 18 items (score 0-72). Higher score indicates high severity.

SECONDARY OUTCOMES:
Proportion of MDS-UPDRS II+III total score change <3 points | 12 weeks
  Proportion of patients whose total score of MDS-UPDRS Ⅱ+Ⅲ changed from baseline by less than 3 points
Movement Disorder Society Unified Parkinson's Disease Rating Scale(MDS-UPDRS)Ⅱ+Ⅲ | 24 weeks
  Part Ⅱ：This measures the motor aspects of activity of daily living and consists of 13 items with scores between 0- 52. Part Ⅲ：This measures the severity of motor symptoms using 18 items (score 0-72). Higher score indicates high severity.
Proportion of MDS-UPDRS II+III total score change <3 points | 24 weeks
  Proportion of patients whose total score of MDS-UPDRS Ⅱ+Ⅲ changed from baseline by less than 3 points
Movement Disorder Society Unified Parkinson's Disease Rating Scale(MDS-UPDRS) part Ⅰ | 12 weeks and 24 weeks
  Assessment of non-motor symptoms of daily life.There are 13 questions, 6 questions in Part 1 A to be completed by the rater and 7 questions in Part 1 B to be completed by the patient.
Cleveland Constipation Score（ CCS），Rome Ⅲ Diagnostic Criteria for Constipation | 12 weeks and 24 weeks
  Constipation improvement was assessed using the Cleveland Constipation Score Change, an 8-question scale with scores ranging from 0 to 30. Evaluate the improvement rate of constipation according to the changes in the proportion of patients who meet the Rome III constipation diagnostic criteria
Parkinson's Disease Sleep Scale-2 (PDSS-2): | 12 weeks and 24 weeks
  Use Parkinson's Disease Sleep Scale-2 (PDSS-2) to assess the patient's sleep improvement. The scale has 15 questions，the higher the score, the worse the sleep.
Clinical Global Impression-severity of illness | 12 weeks and 24 weeks
  Change in scale scores from baseline to assess change in severity of patient's condition
Clinical Global Impression-global improvement | 12 weeks and 24 weeks
  Evaluate the efficacy of patients based on their current condition compared to the time of enrollment
Long-term medication safety | 12 weeks and 24 weeks
  Compare the incidence of adverse reactions between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Houzhen Tuo, PhD, Principal Investigator — Beijing Friendship Hospital
Locations (10):
- China (10):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sampson TR, Debelius JW, Thron T, Janssen S, Shastri GG, Ilhan ZE, Challis C, Schretter CE, Rocha S, Gradinaru V, Chesselet MF, Keshavarzian A, Shannon KM, Krajmalnik-Brown R, Wittung-Stafshede P, Knight R, Mazmanian SK. Gut Microbiota Regulate Motor Deficits and Neuroinflammation in a Model of Parkinson's Disease. Cell. 2016 Dec 1;167(6):1469-1480.e12. doi: 10.1016/j.cell.2016.11.018. PMID 27912057
- [Background] Barichella M, Pacchetti C, Bolliri C, Cassani E, Iorio L, Pusani C, Pinelli G, Privitera G, Cesari I, Faierman SA, Caccialanza R, Pezzoli G, Cereda E. Probiotics and prebiotic fiber for constipation associated with Parkinson disease: An RCT. Neurology. 2016 Sep 20;87(12):1274-80. doi: 10.1212/WNL.0000000000003127. Epub 2016 Aug 19. PMID 27543643
- [Background] Tamtaji OR, Taghizadeh M, Daneshvar Kakhaki R, Kouchaki E, Bahmani F, Borzabadi S, Oryan S, Mafi A, Asemi Z. Clinical and metabolic response to probiotic administration in people with Parkinson's disease: A randomized, double-blind, placebo-controlled trial. Clin Nutr. 2019 Jun;38(3):1031-1035. doi: 10.1016/j.clnu.2018.05.018. Epub 2018 Jun 1. PMID 29891223
- [Background] Kim S, Kwon SH, Kam TI, Panicker N, Karuppagounder SS, Lee S, Lee JH, Kim WR, Kook M, Foss CA, Shen C, Lee H, Kulkarni S, Pasricha PJ, Lee G, Pomper MG, Dawson VL, Dawson TM, Ko HS. Transneuronal Propagation of Pathologic alpha-Synuclein from the Gut to the Brain Models Parkinson's Disease. Neuron. 2019 Aug 21;103(4):627-641.e7. doi: 10.1016/j.neuron.2019.05.035. Epub 2019 Jun 26. PMID 31255487
- [Background] Qian Y, Yang X, Xu S, Wu C, Song Y, Qin N, Chen SD, Xiao Q. Alteration of the fecal microbiota in Chinese patients with Parkinson's disease. Brain Behav Immun. 2018 May;70:194-202. doi: 10.1016/j.bbi.2018.02.016. Epub 2018 Mar 2. PMID 29501802
- [Background] Scheperjans F, Aho V, Pereira PA, Koskinen K, Paulin L, Pekkonen E, Haapaniemi E, Kaakkola S, Eerola-Rautio J, Pohja M, Kinnunen E, Murros K, Auvinen P. Gut microbiota are related to Parkinson's disease and clinical phenotype. Mov Disord. 2015 Mar;30(3):350-8. doi: 10.1002/mds.26069. Epub 2014 Dec 5. PMID 25476529